CLINICAL TRIAL: NCT06765278
Title: Anterior Glenoid Nerve Block Versus Pericapsular Nerve Group (PENG) Block Versus Interscalene Brachial Plexus (ISB) Block for Postoperative Pain Management in Shoulder Arthroscopic Surgeries
Brief Title: Anterior Glenoid Nerve Block Versus Pericapsular Nerve Group Block Versus Interscalene Brachial Plexus Block for Postoperative Pain Management in Shoulder Arthroscopic Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Serry, Assistant Lecturer of Anaesthesia, Intensive Care and Pain Medicine, Faculty of Medicine, Ain Shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD195/2024
Record Dates: First submitted 2024-12-31; First posted 2025-01-09 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Anterior Glenoid Nerve Block; Pericapsular Nerve Group Block; Interscalene Brachial Plexus Block; Postoperative Pain; Shoulder Arthroscopic Surgeries
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interscalene brachial plexus block group (Active Comparator): Patients will receive an Interscalene brachial plexus block.
  Interventions: Other: Interscalene brachial plexus block
- Anterior glenoid nerve block group (Experimental): Patients will receive an anterior glenoid nerve block.
  Interventions: Other: Anterior glenoid nerve block
- Pericapsular nerve group (PENG) block group (Experimental): Patients will receive a pericapsular nerve group (PENG) block.
  Interventions: Other: Pericapsular nerve group block

INTERVENTIONS:
Other: Interscalene brachial plexus block — Patients will receive an Interscalene brachial plexus block.
  Arms: Interscalene brachial plexus block group
Other: Anterior glenoid nerve block — Patients will receive an anterior glenoid nerve block.
  Arms: Anterior glenoid nerve block group
Other: Pericapsular nerve group block — Patients will receive a pericapsular nerve group (PENG) block.
  Arms: Pericapsular nerve group (PENG) block group

SUMMARY:
This study aims to compare between Anterior glenoid nerve block, pericapsular nerve group (PENG) block and Interscalene brachial plexus (ISB) block for post-operative pain management in shoulder arthroscopic surgeries

DETAILED DESCRIPTION:
Major surgeries of the shoulder constitute some of the most commonly performed orthopedic procedures. They often result in moderate to severe postoperative pain thereby requiring a multimodal analgesic approach centered around peripheral nerve blocks.

Postoperative pain management is the part of shoulder surgery to improve patient satisfaction, start rehabilitation process rapidly and decrease for hospital stay.

Interscalene blocks (ISB) are well-studied and established means of providing analgesia following shoulder surgery and are considered the gold standard mode of regional anesthesia and post-operative pain management in shoulder surgeries.

A novel technique: pericapsular nerve group (PENG) block can be effectively and safely applied under ultrasound guidance in shoulder surgery cases for postoperative analgesia. In addition, PENG block targets articular branches with less motor effect compared with interscalene brachial plexus block providing anesthetic and analgesic effect with less complication and better and sooner ambulation.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years.
* No sex predilection.
* American Society of Anesthesiology (ASA) physical status I-II.
* Undergoing shoulder arthroscopic surgeries.

Exclusion Criteria:

* Patient's refusal.
* Patients with a history of drug allergies to study drugs.
* Evidence of local infection at the site of injection.
* Inability to cooperate
* Neuromuscular pathology (example: - Multiple Sclerosis)
* Previous trauma or surgery to the shoulder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to the first dose of pethidine administrated).

SECONDARY OUTCOMES:
Total pethidine consumption | 24 hours postoperatively
  All patients will receive intravenous pethidine (30mg) on demand [Visual Analogue Scale (VAS) score ≥3].
Degree of pain | 24 hours postoperatively
  Degree of pain will be assessed using visual analogue scale (VAS). Each patient will be instructed about postoperative pain assessment with the VAS. VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 6, 12, and 24 hours postoperatively.
Length of hospital stay | Till discharge from hospital (Up to one week).
  Length of hospital stay will be recorded from admission till the discharge from hospital.
Time needed for the patient to freely move the operated limb | Postoperatively (Up to one week).
  Time needed for the patient to freely move the operated limb will be recorded.
Degree of patients satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.